CLINICAL TRIAL: NCT06400017
Title: Mechanism and Application of Deep Brain Stimulation in the Treatment of Parkinson's Disease
Brief Title: Mechanism and Application of DBS in the Treatment of PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Institute of Biotechnology, Academy of Military Medical Sciences, PLA of China (Other); Tsinghua University (Other); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JQ23038-2
Record Dates: First submitted 2024-04-11; First posted 2024-05-06 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Parkinson's Disease and Parkinsonism
Keywords: Cognitive dysfunction; Electrical stimulation of substantia nigra
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: By comparing the behavioral characteristics of the memory paradigm under microelectrode stimulation during DBS operation and the characteristics of the electrophysiological signals behind it, as well as the behavioral characteristics of the memory paradigm under electrical stimulation and the characteristics of brain network activity during DBS startup one month after surgery, we analyzed the regulatory effect of substantia nigra DBS on memory network
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative and One month after the operation microelectrode stimulation of DBS (Experimental): By comparing the behavioral characteristics of the memory paradigm under microelectrode stimulation during DBS operation and the characteristics of the electrophysiological signals behind it, as well as the behavioral characteristics of the memory paradigm under electrical stimulation and the characteristics of brain network activity during DBS startup one month after surgery, we analyzed the regulatory effect of substantia nigra DBS on memory network
  Interventions: Device: microelectrode stimulation of DBS

INTERVENTIONS:
Device: microelectrode stimulation of DBS — Contact selection: According to the electrode position in the image (target reconstruction through CT scan), the electrode located in the substantia nigra is selected as the negative electrode, the contact near the upper part of the substantia nigra is selected as the positive electrode, and the bipolar stimulation mode is selected.
  Stimulation parameters: The frequency was selected as 0/10/130Hz, the pulse width remained unchanged at 90μs, the side effects of patients were observed, and the voltage was slowly increased to 2.0V; The patient voltage was 0 during the spurious stimulation. The washout period was 1 hour

SUMMARY:
Project name: The mechanism and application of deep brain stimulation in the treatment of Parkinson's disease

Objective:

To test the hypothesis that electrical stimulation of substantia nigra regulates cognitive dysfunction in Parkinson's disease and to reveal its electrophysiological mechanism.

Study design:

This study is a self-controlled prospective cohort study. By comparing the behavioral characteristics of the memory paradigm under microelectrode stimulation during DBS operation and the characteristics of the underlying electrophysiological signals, and the behavioral characteristics of the memory paradigm and the characteristics of brain network activity under electrical stimulation when DBS is turned on 1 month after surgery. The regulatory effect of substantia nigra DBS on memory network was analyzed.

Cases: 60

Case selection:

Inclusion criteria:

1)Voluntarily participate in the clinical study and sign the informed consent; 2) Age 50-70 years old, gender unlimited; 3) The clinical diagnosis is consistent with typical PD, and the medical history is less than 20 years; 4) Patients who intend to use 3.0T magnetic resonance compatible dual-channel DBS device (G106R or G106RS, Beijing Pinchi Company) for bilateral subthalamic nucleus DBS surgery to control PD symptoms; 5) MRI excluded patients with obvious structural changes; 6) The visual acuity and hearing of the subjects were basically normal, and the compliance was good, and they could complete the tasks listed in the experimental scheme in accordance with the standards.

Exclusion criteria:

1)Serious mental, cognitive and psychological disorders, unable to sign informed consent or cooperate with the operation and various tasks; 2) There are contraindications for neurosurgery, such as hydrocephalus, cerebral atrophy, cerebrovascular sequelae, heart disease and other cardiovascular and cerebrovascular diseases; 3) There are concomitant diseases that seriously affect health, such as tumors, serious abnormalities of liver and kidney function (indexes more than 3 times normal); 4) There is intracranial space occupation, cerebrovascular disease, mental illness, other neurological diseases, claustrophobia, or there is an implant in the body, which affects the nuclear magnetic scan; 5) The results of the Mini-Mental State Scale (MMSE) <24 or the Montreal Cognitive Assessment Scale (MoCA) <18 in the preoperative assessment, or the results of other scales indicate the presence of severe dementia.

therapeutic schedule： This study did not change the patient's overall treatment regimen, and only electrical stimulation was tested during and after DBS surgery

Efficacy evaluation:

Effectiveness evaluation index (primary efficacy index and secondary efficacy index) : accuracy of memory paradigm, response speed Safety evaluation indicators: blood pressure, heart rate, dual frequency index, patient complaints and symptoms

Statistical methods:

The group t test was used to compare the normal distribution between the measurement data groups. For measurement data with non-normal distribution, Wilcoxon rank sum test was used for comparison between groups.

The study period is January 1, 2024 - December 31, 2026.

DETAILED DESCRIPTION:
Research background The core symptoms of Parkinson's disease (PD) include motor symptoms and non-motor symptoms, among which cognitive dysfunction is the most common and one of the most overlooked non-motor symptoms in patients with advanced PD. Cross-sectional studies have shown that up to 40% of PD patients are combined with cognitive dysfunction at the time of diagnosis, which is manifested by functional decline in memory, executive, attention, language, visuospatial ability and other cognitive subfields. Among them, the memory impairment subtype with episodic memory function decline as the main manifestation is the most common and the fastest progressing. About 10% to 15% of patients with these manifestations will progress to dementia each year, which is four to six times higher than the age-matched non-PD population, and more than 80% of patients with PD will develop dementia within 10 years of diagnosis of PD. This increasing cognitive and memory dysfunction seriously affects the quality of life of patients and the overall treatment effect, often leading to accelerated deterioration of the disease, bringing a heavy burden to the family and society. It can be seen that in-depth exploration of the formation mechanism of PD cognitive and memory dysfunction and the establishment of effective intervention means have become an important proposition to be solved urgently in the field of PD research.

The research group previously tested the behavioral changes of rats in the low frequency electric stimulation group of substantia nigra and the sham stimulation group using behavioral experiments such as nesting experiment and water maze experiment, and found that rats in the low frequency electric stimulation group performed better in the nesting experiment and water maze experiment, suggesting that low frequency electric stimulation of substantia nigra can improve the memory behavioral performance of rats with Parkinson's disease.

The applicant's previous study found that deep brain stimulation (DBS) is an effective means to treat Parkinson's disease, and low frequency electrical stimulation of the substantia nigra can improve episodic memory function in patients with Parkinson's disease. Therefore, the applicant team intends to further study the regulatory effect and mechanism of substantia nigra electrical stimulation on episodic memory, reveal the mechanism of its improvement of cognitive function from the theoretical level, clarify its regulatory effect on cognitive impairment from the technical level, and verify the potential of its treatment of cognitive impairment from the application level, so as to solve the major clinical needs in the diagnosis and treatment of PD cognitive impairment. Bring the Gospel to 5 million PD patients, and help the construction of Beijing International Science and Technology Innovation Center.

Research purpose

1. Main Objective: To verify the hypothesis that electrical stimulation of substantia nigra can regulate cognitive dysfunction in Parkinson's disease, and to reveal its electrophysiological mechanism.
2. Secondary objective: To explore the safety and side effects of electrical stimulation of substantia nigra in regulating cognitive dysfunction.

Research design types, principles and test steps

1. Research design This was a self-controlled prospective cohort study.
2. Sample size and research plan In this study, 60 patients with Parkinson's disease who met the inclusion and exclusion criteria were selected to undergo MRI compatible DBS device implantation. By comparing the behavioral characteristics of the memory paradigm under microelectrode stimulation during DBS operation and the characteristics of the electrophysiological signals behind it, The behavioral characteristics of memory paradigm and brain network activity during electrical stimulation of DBS at 1 month after operation were analyzed, and the regulatory effect of substantia nigra DBS on memory network was analyzed.
3. Study duration January 1, 2024 - December 31, 2026
4. Use DBS equipment and program control 1) DBS equipment manufacturers DBS equipment: dual-channel rechargeable Deep brain stimulation pulse generation System (G106R) compatible with 3.0T magnetic resonance scanning, produced by Beijing Pinchi Medical Equipment Co., LTD.

2) Parameter setting Contact selection: According to the electrode position in the image (target reconstruction through CT scan), the electrode located in the substantia nigra is selected as the negative electrode, the contact near the upper part of the substantia nigra is selected as the positive electrode, and the bipolar stimulation mode is selected.

Stimulation parameters: The frequency was selected as 0/10/130Hz, the pulse width remained unchanged at 90μs, the side effects of patients were observed, and the voltage was slowly increased to 2.0V; The patient voltage was 0 during the spurious stimulation.The washout period was 1 hour.

Side effects: paresthesia, local pain, palpitation, chest tightness, etc. 5. Memory paradigm The episodic memory task paradigm used in this study was designed with the Psychtoolbox (v3.0 version) based on MATLAB2018b(MathWorks, USA). During the operation, the episodic memory paradigm test was conducted 2-3 times for each subject according to the situation, and the total duration of the test was no more than 30 minutes for each subject, or it was stopped at any time according to the subject's will. The paradigm is divided into two phases, in the memory coding phase, 20 silent episodic memory clips (including 10 consecutive event clips and 10 jump event clips) are presented in pseudo-random order. Before each video was played, a cross mark would appear in the center of the screen to remind subjects to look at the center of the screen and reduce eye movement. After each video was played, in order to ensure participants' participation in the passive viewing process, participants were asked to answer questions related to the video (such as determining whether most scenes of the video took place "indoors" or "outdoors"). After the participants memorized and encoded 20 short films, they entered the scene recognition stage. At the beginning of the task, a cross mark appeared in the center of the screen to remind subjects to pay attention to the task, and then scene pictures were displayed (pictures were from 20 films played or not played in the memory coding stage). Subjects were asked to judge whether the scene shown was a selection of short films played in the free memory coding stage. The whole experiment process, the subjects used reactor (RB - 840) answer keys, and the stimulus (video and pictures), and subjects button at the end of your answer by task related electrical synchronizer C - Pod (Cedrus, Us) sends pulses from the experimental computer to Neuro Omega to form time stamps (TTL pulses). Time permitting, the memory encoding and scene recognition phase will be repeated 3-4 times (keeping the same experimental format but replacing it with different experimental clips and test pictures).

Research methods

1. Clinical trials were conducted to verify the regulatory effect of electrical stimulation of substantia nigra under different stimulation modes on episodic memory impairment in PD, and to establish the interdependence between the changes in the firing mode of substantia nigra neurons and the changes in episodic memory function.

1. To evaluate the impact of substantia nigra DBS on episodic memory function of PD subjects: For PD patients to be treated with bilateral subthalaminal nucleus DBS, the cognitive memory function, mental behavior symptoms and daily living ability of the patients were assessed by neuropsychological scale, and those meeting the criteria were selected to be included in the group. The MRI compatible dual-channel DBS device was implanted into the subthalamic nucleus as the target. During the operation, the lowest contact of the DBS electrode was implanted into the substantia nigra according to the electrophysiological signal, and the remaining contact was implanted into the subthalamic nucleus. The position of DBS electrode implantation was reconstructed, and the electrode contacts in or close to the substantia nigra were selected to perform substantia nigra DBS under different parameter combinations such as high frequency and low frequency. Neuropsychological scale was used to evaluate the cognitive memory function of patients, and the influence of substantia nigra DBS under different parameters on the episodic memory function of PD subjects was analyzed. Then to evaluate the effect of substantia nigra DBS on episodic memory function of PD subjects.
2. To study the electrophysiological mechanism of the substantia nigra's participation in episodic memory activities: the experiment of episodic memory task was completed during DBS surgery, and the multi-mode neural electrophysiological signals of brain regions such as substantia nigra, subthalamic nucleus, and dorsolateral prefrontal cortex were recorded synchronously during the process of episodic memory activities, and the behavioral results (accuracy rate, reaction time, etc.) of the completion of the episodic memory tasks were calculated; The dynamic activation/inhibition relationship among the substantia nigra, subthalamic nucleus, dorsolateral prefrontal cortex and other brain regions was analyzed, and the response sequence and dynamic changes of the peak potential, local field potential, and cortical potential under the time-locking relationship were observed, so as to clarify the mutual driving relationship between the brain regions related to episodic memory activities. The activity characteristics of neurons in substantia nigra that respond to episodic memory event boundaries were analyzed, and the relationship between the change of discharge frequency and the formation process of episodic memory events was studied, and the significance of the change of activity on episodic memory events was discussed, so as to analyze the electrophysiological mechanism of various brain regions involved in episodic memory activities.
3. To determine the key time nodes and dose-effect correspondence of the regulation of episodic memory formation by electrical stimulation of substantia nigra: microstimulation or macro stimulation delivered by microelectrode during DBS surgery can be used to predict the effect or side effects of electrical stimulation, and then prepare for the implantation of macro electrode, which is a routine operation in surgery. In this study, the operation of episodic memory paradigm was controlled by programming, and micro-stimulus or macro-stimulus was given before, during and after the presentation of stimuli, respectively, to observe the effects of electrical stimulation with different frequencies, different modes and different stimulation regions on behavioral performance of episodic memory (accuracy rate, reaction time, etc.). To establish the dose-effect correspondence between the relative time node of electrical stimulation, micro-stimulation sites, micro-stimulation parameters and the result of memory formation, and identify the key time node of the regulation of episodic memory formation by electrical stimulation of substantia nigra.

2. Through the study of brain structure and functional connectomics, the optimal stimulus mode and stimulus parameters of substantia nigra DBS regulating episodic memory dysfunction were revealed.

1. The influence of substantia nigra DBS on the functional brain network related to episodic memory was explored by means of functional magnetic resonance imaging (fMRI) technology: the DBS device implanted in this study was an MRI-compatible dual-channel DBS device, and the activity of the brain network could be evaluated by fMRI scanning technology when the device was turned on. In this study, the enrolled patients completed the fMRI scanning of the resting state and the episodic memory task state in the substantia nigra DBS state, calculated the behavioral results (accuracy rate, reaction time, etc.) of the subjects in different groups to complete the episodic memory task, and analyzed the change characteristics and dynamic evolution of the dependent signal of blood oxygen level in the fMRI task state. The brain regions with activation/inhibition of episodic memory task states and their activation/inhibition relationship in time series were analyzed, and the correlation between behavioral results and the characteristics of fMRI signal changes in task states in each group was studied, so as to explore the functional changes of episodic memory brain network before and after substania nigra DBS in PD patients.
2. Verify the results of animal experiments through brain structural connectomics studies, and clarify the correlation between the activated tissue of substantia nigra DBS and the changes in cognitive function: Lead DBS toolkit was used to calculate substantia nigra DBS stimulation-activated tissue volume (VTA) under different parameters, and cognitive behavioral evaluation results under different stimulus parameters were collected, experimental data and patient data of each group were sorted out. The machine learning toolkit was used to analyze the correlation and weight between the changes in behavioral results of the subjects' episodic memory and the subgroups (diagnosis, age, disease course, preoperative evaluation results, imaging indicators, electrophysiological indicators, VTA, fMRI indicators and other information, etc.), so as to clarify the correlation between DBS activated tissue of substantia nigra and the changes in episodic memory function. To search for biomarkers that can predict the changes of episodic memory after DBS, and reveal the optimal stimulation mode and stimulation parameters of substantia nigra DBS in regulating cognitive dysfunction

Concomitant medication Patients will continue to take Parkinson's disease drugs at preoperative dose (or according to the doctor's advice) during perioperative and postoperative periods, and this experiment will not affect the drug usage and dosage of patients.

Observation indicators and inspection time

1. Clinical evaluation: Two evaluations were conducted before surgery and one month after surgery, including the following contents: 1) general information (age, gender, age of onset and course of disease); 2) Drug treatment (drug type, dose, time and side effects); 3) Behavioral assessment: PD patients were evaluated using the Unified Parkinson's Disease Rating Scale(UPDRS) version 3.0; 4) Neuropsychology: In this study, multiple neuropsychological scales will be used for comprehensive assessment of patients, including Mini-mental State Examination (MMSE), the Montreal Cognitive Assessment Scale (MoCA), the Frontal Lobe Function Rating Scale (FAB), the Hamilton Depression Rating Scale for Depression(HRSD), and the Hamilton Anxiety Scale (HRSA).
2. MRI data: 3D T1, T2 axis, T2 crown, BOLD (on and off), DTI sequence. Two times were collected before surgery and one month after surgery.
3. Memory paradigm test data: This project will start the memory paradigm test after the microelectrode enters the substania nigra during the DBS operation, and give electrical stimulation test when some memory stimuli are presented, so as to observe the baseline memory accuracy rate of subjects and the changes in the recognition accuracy rate of new/old objects under the state of electrical stimulation. The memory paradigm test was performed in the ward after surgery to evaluate the cognitive function of the subjects. In addition, when the subjects returned to the hospital one month after the operation, the memory function of the subjects was evaluated with the memory paradigm in the magnetic resonance and fMRI environment, and the changes in the fMRI signal and connectivity of the brain functional areas were observed. Then, the behavioral characteristics of the memory paradigm and the activity characteristics of the brain network under the state of electrical stimulation when DBS was turned on were studied by post-processing analysis technology. The regulatory effect of substantia nigra DBS on memory network was analyzed. We will monitor blood pressure, heart rate, dual-frequency index and other indicators when patients complete the normal form experiment during DBS surgery, and judge whether patients can continue to complete the experiment according to the patient's chief complaint and symptom changes. If all indicators change in a negative direction, the experiment will be terminated timely according to the situation. The safety of using electrical stimulation of substantia nigra to regulate cognitive function was evaluated according to the changes of blood pressure, heart rate, dual frequency index, complaints and symptoms of patients after completing the normal form experiment.

Follow-up time Follow-up will be completed at DBS startup 1 month after surgery.

Clinical evaluation

1. Efficacy evaluation: Changes in the corresponding clinical scales of patients at each follow-up point are shown in observation indicators and examination time.
2. Safety evaluation: Adverse events were described by the number of adverse events and the incidence rate, and the incidence rate was tested for significance between groups. At the same time, the specific manifestation, degree and relationship between all adverse events and devices were described in detail. Including surgery-related adverse reactions, stimulus-related adverse reactions and device-related adverse reactions.

Known and potential risks and benefits of the project, as well as risk disposal plans This study will require you to complete a cognitive function test during the operation, which requires only a simple operation of the keyplate and lasts about 20-30 minutes, during which the operation will be stopped and the surgical incision will be covered with a sterile towel. Previous studies done in our center and other centers have shown that this testing procedure does not significantly increase the degree of infection of the incision. Nor does it significantly increase the overall risk of surgery; In part of the testing process, we will use a micro-current below 50uA for electrical stimulation, which is not substantially different from the electrical stimulation used to test the efficacy of surgery, and the intensity is significantly weaker than the efficacy test current. Previous studies have not found that such intensity of the current will induce epilepsy, bleeding, necrosis and other complications, and the subjects have not reported obvious subjective discomfort. About 1 month after surgery, when you participate in the follow-up, a professional program control physician will test the changes in cognitive function under electrical stimulation of the substantia nigra. The parameters of electrical stimulation used in the process are within the safe range of parameters, usually without significant discomfort, and the effects of electrical stimulation disappear immediately after the stimulator is turned off.

Considering that participation in this study will require the cooperation of patients during and after the operation, and may lead to a slight extension of the operation time, and the need for post-operation debugging and corresponding inspection, the project team will cooperate with Beijing Pinchi Medical Equipment Co., Ltd. to provide further support and follow-up services for patients.

In addition, patients will return to the hospital about 1 month after surgery for a free head MRI and fMRI scan, as well as a detailed brain evaluation and examination. In addition, we will also provide a transportation subsidy of 400 yuan for patients.

Data preservation The researchers established an independent study number for each subject, named the corresponding data with the study number, and deleted the patient name and hospital number information from all the data. The study data included behavioral data in.mat format, CT and MRI data in.dcm format, EEG data in.mpx format and image data in.mp4 format. Keep the original data for 10 years after the completion or termination of the study.

Data security inspection Data and safety monitors were set up in this study, all adverse events were recorded in detail, properly handled and tracked until properly resolved or the disease was stable, and serious adverse events and unexpected events were reported to the ethics Committee, competent authorities, sponsors and drug regulatory authorities in a timely manner in accordance with relevant systems; The principal investigator conducts a cumulative review of all adverse events on a regular basis, and investigator meetings are convened when necessary to assess the risks and benefits of the study.

Statistical processing SPSS 22.0 software or SAS9.4 were used for analysis. In bilateral tests, P < 0.05 was considered to have significant differences. Measurement data were described by mean, standard deviation, maximum, minimum, median, 25th and 75th quantile. Group t test was used to compare the normal distribution measurement data among groups. For measurement data with non-normal distribution, Wilcoxon Rank Sum test was used for inter-group comparison.

Ethical considerations Recruitment will be conducted in the Clinical Trial Office of Functional Neurosurgery at Tiantan Hospital, and we will endeavour to ensure a closed environment to protect the privacy of the subjects. In order to obtain informed consent from the subjects and their families, we will provide written materials in non-technical terms to help them better understand the study content. We will ensure that participants and their families have sufficient time to consider whether to participate in the study and that they are aware of their right to withdraw from the study at any time. After subjects express their willingness to participate in the study, we will require them to sign a written informed consent as an official proof of participation in the clinical study. This informed consent form will be kept safe for review as part of the clinical study documentation.

During the course of the study, we will strictly protect the subject's personal information to ensure that it will not be disclosed to any unauthorized third party. We will take various measures, including but not limited to data encryption, access control, etc., to ensure that subjects' privacy is adequately protected.

In addition, we will try to avoid any undue influence on the subject. We will avoid providing an informed notification hours before the procedure to ensure that the subject has sufficient time to consider and prepare. We will also avoid being informed by well-known experts in person to avoid excessive psychological pressure on the subjects. For older patients of the investigator, we will ask another researcher or student to inform them on behalf of the investigator to avoid possible conflicts of interest. At the same time, we will also avoid including students or subordinates of the researcher in the research object, so as to ensure the fairness and objectivity of the research.

We will strictly follow the regulatory requirements to ensure that the research process is legal and compliant, and that the rights and interests of the subjects are fully protected. We will carry out this study with a good faith and responsible attitude, aiming to provide new ideas and methods for the treatment of Parkinson's disease, and bring better treatment results and quality of life for patients.

Confidentiality of information The subjects' medical information will be combined and used to study treatments. All information will be coded and will not contain the subject's name or any other information that directly identifies the subject. Information that is not relevant to the study (such as information about previous illnesses, infectious disease history) will not be provided to other parties.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the clinical study and sign the informed consent;
* Age 50-70 years old, gender unlimited;
* The clinical diagnosis is consistent with typical PD, and the medical history is less than 20 years;
* Patients who intend to use 3.0T magnetic resonance compatible dual-channel DBS device (G106R or G106RS, Beijing Pinchi Company) for bilateral subthalamic nucleus DBS surgery to control PD symptoms;
* MRI excluded patients with obvious structural changes;
* The visual acuity and hearing of the subjects were basically normal, and the compliance was good, and they could complete the tasks listed in the experimental scheme in accordance with the standards.

Exclusion Criteria:

* Serious mental, cognitive and psychological disorders, unable to sign informed consent or cooperate with the operation and various tasks;
* There are contraindications for neurosurgery, such as hydrocephalus, cerebral atrophy, cerebrovascular sequelae, heart disease and other cardiovascular and cerebrovascular diseases;
* There are concomitant diseases that seriously affect health, such as tumors, serious abnormalities of liver and kidney function (indexes more than 3 times normal);
* There is intracranial space occupation, cerebrovascular disease, mental illness, other neurological diseases, claustrophobia, or there is an implant in the body, which affects the nuclear magnetic scan;
* The results of the Mini-Mental State Scale (MMSE) <24 or the Montreal Cognitive Assessment Scale (MoCA) <18 in the preoperative assessment, or the results of other scales indicate the presence of severe dementia.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in recognition accuracy of new/old objects between baseline and under electrical stimulation | From the middle of DBS surgery to one month after surgery
  In this project, after the microelectrode was inserted into the substantia nigra during DBS surgery, the memory paradigm test was started, and some memory stimuli were presented with electrical stimulation test at the same time, so as to observe the baseline memory accuracy of the subjects and the changes in the recognition accuracy of new/old objects under the state of electrical stimulation. The memory paradigm test was performed in the ward after surgery to evaluate the cognitive function of the subjects
Changes of fMRI signal and connectivity in brain functional areas | From preoperative to one month postoperative
  In this study, SPM12 and DPABI were used to preprocess the resting-state fMRI data and calculate the functional connectivity, locate the location of the dorsolateral prefrontal lobe, establish the resting-state brain network between the substantia nigra and the dorsolateral prefrontal lobe, calculate the functional connectivity between the substantia nigra and the dorsolateral prefrontal lobe, and design the surgical path. The maximum functional connectivity between the dorsolateral prefrontal cortex, substantia nigra and subthalamic nucleus was calculated according to the results of resting-state fMRI. All subjects underwent 7.0T and 3.0T MR Scans before and after surgery, respectively. Scanning sequences included 3D-T1-weighted images, axial coronal T2-weighted images, 3D-Flair sequences, etc. In addition, all participants completed the resting-state and task-state fMRI scans before and after the operation, and the post-operation task-state fMRI scan was performed with DBS on
Multimode neuroelectrophysiological signal recording | During DBS surgery
  In this study, the spike potential and local field potential signals at the location of the microelectrode tip were recorded simultaneously, and the cortical potential signals of the dorsolateral prefrontal cortex were collected by a custom-made ring electrode to analyze the spatio-temporal characteristics of the SN and the dorsolateral prefrontal cortex during the formation of episodic memory encoding. The microelectrode recorded microvolt electrophysiological signals within 0.2-0.3mm around the microelectrode. The macroelectrode recorded the surrounding local field potential signal. In this way, the spike potential signal and local field potential signal at the tip of the microelectrode, the local field potential signal 3mm behind the tip, and the cortical potential signal could be recorded synchronously.
Mini-mental State Examination Score | From preoperative to one month postoperative
  The DBS device was implanted at the subthalamic nucleus. According to the electrophysiological signal during the operation, the lowest contact of the DBS electrode was implanted into the substantia nigra, and the remaining contacts were implanted into the subthalamic nucleus. The cognitive memory function of the patients was assessed by Mini-mental State Examination before surgery, and then the cognitive memory function of the patients in no stimulation, low frequency and high frequency substantia nigra DBS states was assessed by Mini-mental State Examination Score one month after surgery. The effects of substantia nigra DBS with different parameters on the memory function of PD subjects were analyzed. The scale has a minimum value of 0 and a maximum value of 30, with higher scores indicating better outcomes.
Montreal Cognitive Assessment Score | From preoperative to one month postoperative
  The DBS device was implanted at the subthalamic nucleus. According to the electrophysiological signal during the operation, the lowest contact of the DBS electrode was implanted into the substantia nigra, and the remaining contacts were implanted into the subthalamic nucleus. The cognitive memory function of the patients was assessed by Montreal Cognitive Assessment before surgery, and then the cognitive memory function of the patients in no stimulation, low frequency and high frequency substantia nigra DBS states was assessed by Montreal Cognitive Assessment one month after surgery. The effects of substantia nigra DBS with different parameters on the memory function of PD subjects were analyzed. The scale has a minimum value of 0 and a maximum value of 30, with higher scores indicating better outcomes.
Frontal Lobe Function Rating Scale | From preoperative to one month postoperative
  The DBS device was implanted at the subthalamic nucleus. According to the electrophysiological signal during the operation, the lowest contact of the DBS electrode was implanted into the substantia nigra, and the remaining contacts were implanted into the subthalamic nucleus. The cognitive memory function of the patients was assessed by Frontal Lobe Function Rating Scale before surgery, and then the cognitive memory function of the patients in no stimulation, low frequency and high frequency substantia nigra DBS states was assessed by Frontal Lobe Function Rating Scale one month after surgery. The effects of substantia nigra DBS with different parameters on the memory function of PD subjects were analyzed. The scale has a minimum value of 0 and a maximum value of 18, with higher scores indicating better outcomes.
Trail Making Test Time | From preoperative to one month postoperative
  The DBS device was implanted at the subthalamic nucleus. According to the electrophysiological signal during the operation, the lowest contact of the DBS electrode was implanted into the substantia nigra, and the remaining contacts were implanted into the subthalamic nucleus. The cognitive memory function of the patients was assessed by Trail Making Test before surgery, and then the cognitive memory function of the patients in no stimulation, low frequency and high frequency substantia nigra DBS states was assessed by Trail Making Test Time one month after surgery. The effects of substantia nigra DBS with different parameters on the memory function of PD subjects were analyzed. The scale has a minimum value of 0 and a maximum value of 300, with higher scores indicating worse outcomes.
Auditory Verbal Learning Test | From preoperative to one month postoperative
  The DBS device was implanted at the subthalamic nucleus. According to the electrophysiological signal during the operation, the lowest contact of the DBS electrode was implanted into the substantia nigra, and the remaining contacts were implanted into the subthalamic nucleus. The cognitive memory function of the patients was assessed by Auditory Verbal Learning Test before surgery, and then the cognitive memory function of the patients in no stimulation, low frequency and high frequency substantia nigra DBS states was assessed by Auditory Verbal Learning Test Score one month after surgery. The effects of substantia nigra DBS with different parameters on the memory function of PD subjects were analyzed. The scale has a minimum value of 0 and a maximum value of 24, with higher scores indicating better outcomes.
Digital Span Test | From preoperative to one month postoperative
  The DBS device was implanted at the subthalamic nucleus. According to the electrophysiological signal during the operation, the lowest contact of the DBS electrode was implanted into the substantia nigra, and the remaining contacts were implanted into the subthalamic nucleus. The cognitive memory function of the patients was assessed by Digital Span Test before surgery, and then the cognitive memory function of the patients in no stimulation, low frequency and high frequency substantia nigra DBS states was assessed by Digital Span Test Score one month after surgery. The effects of substantia nigra DBS with different parameters on the memory function of PD subjects were analyzed. The scale has a minimum value of 5 and a maximum value of 22, with higher scores indicating better outcomes.
Digital Order Test | From preoperative to one month postoperative
  The DBS device was implanted at the subthalamic nucleus. According to the electrophysiological signal during the operation, the lowest contact of the DBS electrode was implanted into the substantia nigra, and the remaining contacts were implanted into the subthalamic nucleus. The cognitive memory function of the patients was assessed by Digital Order Test before surgery, and then the cognitive memory function of the patients in no stimulation, low frequency and high frequency substantia nigra DBS states was assessed by Digital Order Test Score one month after surgery. The effects of substantia nigra DBS with different parameters on the memory function of PD subjects were analyzed. The scale has a minimum value of 0 and a maximum value of 12, with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: lin shi, M.D., Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China